CLINICAL TRIAL: NCT02761733
Title: Researching the Effectiveness of a Decision-Support Tool for Adult Consumers With Mental Health Needs and Their Care Managers
Brief Title: The Effectiveness of a Decision-Support Tool for Adult Consumers With Mental Health Needs and Their Care Managers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Felton Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CE-12-11-4309
Record Dates: First submitted 2016-01-20; First posted 2016-05-04 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Mental Disorders
Keywords: Shared Decision Making; Case Management; Decision Aid
MeSH Terms: conditions — Mental Disorders | interventions — Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mPOWR System (Experimental): Moving Patient Outcomes toward Wellness and Recovery (mPOWR) consists of an assessment questionnaire and decision support tools which map onto 6 life domains which are measured by the questionnaire.
  Interventions: Behavioral: Moving Patient Outcomes toward Wellness and Recovery (mPOWR)
- Control (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Moving Patient Outcomes toward Wellness and Recovery (mPOWR) — An mPOWR intervention and toolkit that consists of strategies, prompts, and decision aids designed to foster patient involvement in treatment. The mPOWR intervention includes a questionnaire that assesses quality of life and consumer functioning for use in the development of consumer-centered goals and outcomes within the mPOWR intervention.
  Arms: mPOWR System

SUMMARY:
The primary goal of the proposed study is to investigate the implementation and effectiveness of the mPOWR (Moving Patient-centered Outcomes through Wellness and Recovery) in diverse urban and rural community mental health settings. The study compares patient participation and outcomes using the mPOWR system to a usual care control condition. Four community mental health agencies participate in the research: two in San Francisco (urban) and two in N.M. (rural). One site in each setting serves as the mPOWR implementation site and the other serves as the control site. Service sites were randomly assigned to intervention or usual care conditions. A quasi experimental design was used; only eligible participants were enrolled in the study (e.g., exclusion criteria of moderate to severe cognitive impairment, patient services structured for provision of mPOWR implementation, etc.). The study design will employ repeated quantitative measures to assess change in outcomes within and across conditions over time. Qualitative methods in the form of focus group interviews will also be used to round out the information obtained about patient and provider expectations and experiences. Primary outcomes of interest include: Short Form Health Survey-12 (SF-12; physical and mental health aspects of health and well-being); Outcome Rating Scale (ORS; general well-being, personal well-being, close relationships, and work/school/friend relationships); Shared Decision Making Questionnaire (congruence of patient's and provider's participation in therapeutic decision making and patient's understanding of treatment and treatment options); Working Alliance Inventory (perception of therapeutic alliance); and Satisfaction Questionnaire (communication patterns between physicians and their patients).

DETAILED DESCRIPTION:
Research on the impact of decision-support tools for providers and patients has not included frontline care managers within community mental health settings. In particular, the care management field lacks effective models for integrating results-based and patient-centered care into routine practice with diverse adults with complex mental health and social service needs. For over five years, Family Service Agency of San Francisco (FSA) developed and piloted a mental health decision-support tool entitled the Assessment Diagnostic Evaluation and Planning Tool (ADEPT) for use by patients and front-line providers. The ADEPT was developed by a team of researchers, frontline providers, and FSA patients to collect data and track patient progress over time. Yet, its strong focus on diagnostic screening and excessive length limited its relevance to patients in guiding service decisions. Over the past two years, a team of FSA patients and care managers revised the tool, eliminating its diagnostic component and retaining two measures of quality of life and community living skills that were reviewed and/or adapted by patients to reflect meaningful outcomes in the delivery of services. Decision aids and a communications toolkit were also developed to support the use of shared-decision making (SDM) processes in the provision of services. Together, these instruments and tools make up the Moving Patient Outcomes toward Wellness and Recovery (mPOWR) system. mPOWR ensures that the patient-provider relationship remains focused on patient identified outcomes and use of SDM throughout care. The primary goal of the study is to investigate the implementation and effectiveness of the mPOWR in diverse urban and rural community mental health settings.

FSA has partnered with senior faculty from the University of New Mexico to serve as independent researchers for this study. The study involves four community mental health agencies: two in San Francisco (urban) and two in N.M. (rural). One (randomly chosen) site in each setting serves as the mPOWR implementation site and the other serves as the control site. The study population initially enrolled included 240 (60/site X 4 sites) diverse adults with chronic mental health conditions. The specific aims for this study are: (1) To improve patient and provider participation in shared-decision making and engagement in mental health treatment, to improve [patient] personal Quality of Life, and to improve [patient] access to community/social services; (2) To increase patient understanding of their treatment and of treatment options; to increase their personal treatment progress; (3) To increase patient functionality and sense of perceived support for their therapeutic outcomes.

Primary outcomes of interest include: Short Form Health Survey-12 (SF-12; physical and mental health aspects of health and well-being); Outcome Rating Scale (ORS; general well-being, personal well-being, close relationships, and work/school/friend relationships); Shared Decision Making Questionnaire (congruence of patient's and provider's participation in therapeutic decision making and patient's understanding of treatment and treatment options); Working Alliance Inventory (perception of therapeutic alliance); and Satisfaction Questionnaire (communication patterns between physicians and their patients). Qualitative methods in the form of focus group interviews will also be used to round out the information obtained about patient and provider expectations and experiences. Data will be collected in a time series design.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18 who are receiving mental health services.

Exclusion Criteria:

Temporary Exclusion:

* Disruptive, aggressive, or severely disorganized behaviors;
* Visibly intoxicated or under the influence of illicit drugs.

General Exclusion:

* Moderate to severe cognitive impairment;
* Developmental disability that precludes comprehension;
* Language issues: Intervention is only offered in English and Chinese;
* Patient services structured for provision of mPOWR implementation (e.g., not in and out of inpatient or crisis stabilization services).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Chu, PhD, Principal Investigator — Felton Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larson CO, Schlundt D, Patel K, Beard K, Hargreaves M. Validity of the SF-12 for use in a low-income African American community-based research initiative (REACH 2010). Prev Chronic Dis. 2008 Apr;5(2):A44. Epub 2008 Mar 15. PMID 18341779
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Johnson JA, Coons SJ. Comparison of the EQ-5D and SF-12 in an adult US sample. Qual Life Res. 1998 Feb;7(2):155-66. doi: 10.1023/a:1008809610703. PMID 9523497
- [Background] Miller, S., et al., The Outcome Rating Scale: A Preliminary Study of the Reliability, Validity, and Feasibility of a Brief Visual Analog Measure. J Brief Therapy, 2003. 2(2): p. 91-100.
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Hanson, W., K. Curry, and D. Bandalos, Reliability Generalization of Working Alliance Inventory Scale Scores. Educational and Psychological Measurement, 2002. 62(4): p. 659-673.
- [Background] Horvath, A. and L. Greenberg, Development and validation of the Working Alliance Inventory. J Counseling Psychology, 1989. 36: p. 223-233.
- [Background] Campbell C, Lockyer J, Laidlaw T, Macleod H. Assessment of a matched-pair instrument to examine doctor-patient communication skills in practising doctors. Med Educ. 2007 Feb;41(2):123-9. doi: 10.1111/j.1365-2929.2006.02657.x. PMID 17269944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The research team distributed recruitment letters (in English and Chinese) via mail and in person in all four research sites. With assistance from case managers, research assistants introduced themselves to patients and invited participation. Recruitment occurred from October 2013 to June 2014.
Pre-assignment Details: Enrollment was not directly related to the assignment of intervention, which was randomized at the site level. The screening predetermined criteria (exclusion of cognitive impairment). The number of individuals found eligible to participate was 266, and the research team subsequently randomly selected 240 participants.
Groups:
- Intervention Site - Urban Setting: The clinical case mangers at this site were trained to implement the intervention. This site is based in inner city San Francisco, CA. (Geriatric Services West)
- Control Site - Urban Setting: Treatment as usual. This site is based in inner city San Francisco, CA. (Gough Street Clinic)
- Intervention Site - Rural Setting: The clinical case mangers at this site were trained to implement the intervention. This site is based in rural New Mexico. (Tri-County Community Services in Taos, NM)
- Control Site - Rural Setting: Treatment as usual. This site is based in rural New Mexico. (Mental Health Resources in Clovis, NM)
Period: Overall Study
Arm/Group | Intervention Site - Urban Setting | Control Site - Urban Setting | Intervention Site - Rural Setting | Control Site - Rural Setting
Started | 60 | 60 | 60 | 60
9/30/2014 (Completion of the 2nd Wave of Data Collection) | 53 | 56 | 48 | 55
3/31/2015 (Completion of the 3rd Wave of Data Collection) | 48 | 47 | 43 | 50
9/30/2015 (Completion of the 4th Wave of Data Collection) | 40 | 44 | 33 | 50
Completed | 30 | 39 | 33 | 45
Not Completed | 30 | 21 | 27 | 15
Not completed — Death | 3 | 5 | 1 | 1
Not completed — Lost to Follow-up | 6 | 7 | 0 | 3
Not completed — Physician Decision | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Discharged from Study Site | 10 | 9 | 25 | 11
Not completed — Cognitive Impairment | 5 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Site - Urban Setting | Control Site - Urban Setting | Intervention Site - Rural Setting | Control Site - Rural Setting | Total
Number analyzed (Participants) | 60 | 60 | 60 | 60 | 240
Age, Categorical [Count of Participants; unit: Participants] — Population: Two clients at the rural control site did not report demographic data.
  Participants
    number analyzed (Participants) | 60 | 60 | 60 | 58 | 238
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 13 | 19 | 54 | 50 | 136
    >=65 years | 47 | 41 | 6 | 8 | 102
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 34 | 30 | 28 | 35 | 127
  Male | 26 | 29 | 32 | 25 | 112
  Other | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White, not Hispanic | 30 | 38 | 25 | 37 | 130
  Race/Ethnicity: Black, not Hispanic | 6 | 10 | 0 | 0 | 16
  Race/Ethnicity: Hispanic | 5 | 4 | 32 | 20 | 61
  Race/Ethnicity: Asian or Pacific Islander | 16 | 5 | 0 | 0 | 21
  Race/Ethnicity: American Indian or Alaskan Native | 0 | 1 | 1 | 0 | 2
  Race/Ethnicity: Mixed | 0 | 1 | 0 | 0 | 1
  Race/Ethnicity: Other | 3 | 1 | 1 | 0 | 5
  Race/Ethnicity: Unknown | 0 | 0 | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 60 | 60 | 60 | 240

OUTCOME MEASURES:

1. Primary Outcome: Short Form Health Survey-12 (SF-12), Physical Symptoms Subscale
Description: The physical health subscale (PCS-12; Physical Component Summary) of the SF-12 (Health Survey Short Form-12) was utilized in the current study to assess physical aspects of health and well-being48. The measure includes twelve questions asking about overall health, limitations from health conditions, physical health, emotional well-being and daily activities, and feelings over the past four weeks, utilizing variable Likert scale response choice options. The aggregate PCS subscale score of the SF-12 is calculated utilizing norm-based scoring with a weighted sum (Ware, Kosinski, & Keller, 1995). PCS scores in the present study ranged from 13.2 to 65.6, with higher values indicating better physical health.
Time Frame: Change in scores on the SF-12 from Baseline to 24 month follow-up
Population: Several factors influenced variability in the number of participants analyzed across time points. First, patients may have responded to some items but opted out of others because of questionnaire length or comprehension considerations. Second, some patients were available at baseline but were unavailable at subsequent time points, or vice versa.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Site - Urban Setting | Control Site - Urban Setting | Intervention Site - Rural Setting | Control Site - Rural Setting
Number analyzed (Participants) | 60 | 60 | 60 | 60
units on a scale
  Baseline: number analyzed (Participants) | 46 | 55 | 58 | 59
  Baseline | 38.167 (11.067) | 38.601 (10.595) | 37.187 (12.585) | 37.108 (10.148)
  24 Month Follow-up: number analyzed (Participants) | 29 | 30 | 32 | 45
  24 Month Follow-up | 34.386 (8.801) | 35.884 (12.343) | 36.354 (9.734) | 37.163 (12.555)
Statistical Analysis 1: Comparison: Intervention Site - Urban Setting; Test type: Superiority or Other; p = .0679, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -3.3652, 95% CI 2-sided [-6.9559 to .2255] — Satterthwaite adjusted df = 173
Statistical Analysis 2: Comparison: Control Site - Urban Setting; Test type: Superiority or Other; p = .0999, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -2.8820, 95% CI 2-sided [-6.2957 to 0.5317] — Satterthwaite adjusted df = 165
Statistical Analysis 3: Comparison: Intervention Site - Rural Setting; Test type: Superiority or Other; p = .5588, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -1.0139, 95% CI 2-sided [-4.4957 to 2.3779] — Satterthwaite adjusted df = 148
Statistical Analysis 4: Comparison: Control Site - Rural Setting; Test type: Superiority or Other; p = .8532, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = .2798, 95% CI 2-sided [-2.6771 to 3.2367] — Satterthwaite adjusted df = 136

2. Primary Outcome: Short Form Health Survey-12 (SF-12) Mental Symptoms
Description: The mental health subscale (MCS-12; Mental Component Summary) of the SF-12 (Health Survey Short Form-12) was utilized in the current study to assess mental aspects of health and well-being48. The measure includes twelve questions asking about overall health, limitations from health conditions, physical health, emotional well-being and daily activities, and feelings over the past four weeks, utilizing variable Likert scale response choice options. The physical health subscale of the SF-12 was utilized as a key client functioning outcome in the current study. The aggregate MCS subscale score of the SF-12 is calculated utilizing norm-based scoring with a weighted sum (Ware, Kosinski, & Keller, 1995). MCS scores in the present study ranged from 9.6 to 72.0, with higher values indicating better physical health.
Time Frame: Change in scores on the SF-12 from Baseline to 24 month follow-up Description: The Health Survey Short Form-12 (SF-12) includes 12 items that assess for physical and mental aspects of health and well-being.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Site - Urban Setting | Control Site - Urban Setting | Intervention Site - Rural Setting | Control Site - Rural Setting
Number analyzed (Participants) | 60 | 60 | 60 | 60
units on a scale
  Baseline: number analyzed (Participants) | 46 | 55 | 58 | 59
  Baseline | 43.828 (14.150) | 38.647 (13.623) | 34.153 (12.288) | 39.970 (13.033)
  24 Month Follow-up: number analyzed (Participants) | 29 | 30 | 32 | 45
  24 Month Follow-up | 39.931 (12.795) | 39.570 (13.714) | 35.850 (11.915) | 37.768 (11.092)
Statistical Analysis 1: Comparison: Intervention Site - Urban Setting; Test type: Superiority or Other; p = .0988, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -3.4524, 95% CI 2-sided [-7.5302 to 0.6254] — Satterthwaite adjusted df = 180
Statistical Analysis 2: Comparison: Control Site - Urban Setting; Test type: Superiority or Other; p = .8760, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -.3087, 95% CI 2-sided [-4.1799 to 3.5625] — Satterthwaite adjusted df = 166
Statistical Analysis 3: Comparison: Intervention Site - Rural Setting; Test type: Superiority or Other; p = .1878, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = 2.541, 95% CI 2-sided [-1.2234 to 6.3054] — Satterthwaite adjusted df = 153
Statistical Analysis 4: Comparison: Control Site - Rural Setting; Test type: Superiority or Other; p = .3330, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -1.6237, 95% CI 2-sided [-4.9000 to 1.6526] — Satterthwaite adjusted df = 143

3. Primary Outcome: Outcome Rating Scale (ORS)
Description: The Outcome Rating Scale (ORS) was utilized as a repeated measure of general therapy outcomes and quality of life changes during the course of therapy. The Outcome Rating Scale includes a visual analog scale (a horizontal line on which the participants marks how well they are doing within the last week from low to high) that records four questions about general well-being, personal well-being, close relationships, and work/school/friend relationships. Physical marks for each of four domains on the visual analog scale are measured by research team members with a ruler and converted to a score from 1 to 100. The four items are then averaged for an overall therapy outcome score. The total averaged ORS score ranges from 1 to 100, with higher scores indicating a better outcome. Analyses will examine treatment progress via change in ORS scores from pre- to post-intervention.
Time Frame: Change in scores on the Outcome Rating Scale from Baseline to 24 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Site - Urban Setting | Control Site - Urban Setting | Intervention Site - Rural Setting | Control Site - Rural Setting
Number analyzed (Participants) | 60 | 60 | 60 | 60
units on a scale
  Baseline: number analyzed (Participants) | 58 | 59 | 60 | 60
  Baseline | 58.085 (24.192) | 49.003 (29.995) | 57.522 (23.978) | 59.583 (24.171)
  24 Month Follow-up: number analyzed (Participants) | 30 | 39 | 33 | 45
  24 Month Follow-up | 54.083 (29.634) | 56.987 (28.737) | 47.083 (29.460) | 61.433 (21.688)
Statistical Analysis 1: Comparison: Intervention Site - Urban Setting; Test type: Superiority or Other; p = .6588, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -1.9284, 95% CI 2-sided [-10.4728 to 6.6160] — Satterthwaite adjusted df = 175
Statistical Analysis 2: Comparison: Control Site - Urban Setting; a priori test; Test type: Superiority or Other; p = .2633, Mixed Models Analysis — Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Satterthwaite adjusted df = 169; Mean Difference (Net) = 4.3959, 95% CI 2-sided [-2.2237 to 11.0155]
Statistical Analysis 3: Comparison: Intervention Site - Rural Setting; a priori test; Test type: Superiority or Other; p = .0343, Mixed Models Analysis — Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Satterthwaite adjusted df = 166; Mean Difference (Net) = -8.9703, 95% CI 2-sided [-17.2107 to -0.7299] — Satterthwaite adjusted df = 166
Statistical Analysis 4: Comparison: Control Site - Rural Setting; a priori test; Test type: Superiority or Other; p = .3126, Mixed Models Analysis — Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = 3.7297, 95% CI 2-sided [-3.4864 to 10.9458] — Satterthwaite adjusted df = 163

4. Primary Outcome: Shared Decision Making Questionnaire
Description: A 6-item modified version of the Shared Decision Making Questionnaire (SDM-Q-9) 46 was utilized to assess client reports about the degree to which their provider involved them in understanding and making a treatment decision. Examples items included "My provider discussed the advantages and disadvantages of options and strategies" or "My provider helped me understand all the information" measured on a 6-point scale (completely disagree, strongly disagree, somewhat disagree, somewhat agree, strongly agree, and completely agree). The total average score ranges from 1 to 6 with higher scores indicating a better outcome of greater shared decision making. Analyses will examine change in Shared Decision Making Questionnaire scores from pre- to post-intervention.
Time Frame: Change in scores on the Shared Decision Making Questionnaire from Baseline to 24 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Site - Urban Setting | Control Site - Urban Setting | Intervention Site - Rural Setting | Control Site - Rural Setting
Number analyzed (Participants) | 60 | 60 | 60 | 60
units on a scale
  Baseline: number analyzed (Participants) | 37 | 33 | 47 | 40
  Baseline | 4.698 (1.289) | 4.005 (1.293) | 4.995 (0.907) | 5.220 (0.673)
  24 Month Follow-up: number analyzed (Participants) | 21 | 25 | 29 | 36
  24 Month Follow-up | 4.512 (0.872) | 4.363 (0.999) | 5.270 (0.827) | 5.239 (0.665)
Statistical Analysis 1: Comparison: Intervention Site - Urban Setting; Test type: Superiority or Other; p = .5840, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -.1241, 95% CI 2-sided [-.5675 to .3193] — Satterthwaite adjusted df = 142
Statistical Analysis 2: Comparison: Control Site - Urban Setting; Test type: Superiority or Other; p = .2404, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = .2642, 95% CI 2-sided [-.1754 to .7038] — Satterthwaite adjusted df = 184
Statistical Analysis 3: Comparison: Intervention Site - Rural Setting; Test type: Superiority or Other; p = .1074, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = .3192, 95% CI 2-sided [-.0667 to .7051] — Satterthwaite adjusted df = 129
Statistical Analysis 4: Comparison: Control Site - Rural Setting; Test type: Superiority or Other; p = .7677, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = .0576, 95% CI 2-sided [-.3238 to .4390] — Satterthwaite adjusted df = 131

5. Primary Outcome: Working Alliance Inventory
Description: The Working Alliance Inventory measures the perception of therapeutic alliance in a clinical dyad during the process of developing a relationship required for effective psychotherapy. The current study utilized the client version of the Working Alliance Inventory included 7 items measured on a 7-point scale (never, rarely, occasionally, sometimes, often, very often, always). Example items included "I am confident in my provider's ability to help me" and "My provider and I trust one another." The Working Alliance Inventory total average score ranges from 1 to 7, with high scores indicating a more positive outcome. Analyses will examine change in patient-reported Working Alliance Inventory scores from pre- to post-intervention.
Time Frame: Change in scores on the Working Alliance Inventory from Baseline to 24 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Site - Urban Setting | Control Site - Urban Setting | Intervention Site - Rural Setting | Control Site - Rural Setting
Number analyzed (Participants) | 60 | 60 | 60 | 60
units on a scale
  Baseline: number analyzed (Participants) | 54 | 58 | 60 | 60
  Baseline | 5.896 (1.065) | 5.494 (1.086) | 6.203 (0.751) | 6.058 (1.045)
  24 Month Follow-up: number analyzed (Participants) | 29 | 37 | 34 | 46
  24 Month Follow-up | 5.842 (0.941) | 5.810 (1.344) | 5.723 (1.182) | 5.751 (1.042)
Statistical Analysis 1: Comparison: Intervention Site - Urban Setting; Test type: Superiority or Other; p = .9046, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -.0260, 95% CI 2-sided [-.4507 to .3987] — Satterthwaite adjusted df = 182
Statistical Analysis 2: Comparison: Control Site - Urban Setting; Test type: Superiority or Other; p = .2518, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = .2258, 95% CI 2-sided [-.1591 to .6107] — Satterthwaite adjusted df = 173
Statistical Analysis 3: Comparison: Intervention Site - Rural Setting; Test type: Superiority or Other; p = .0338, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -.4370, 95% CI 2-sided [-.8370 to -.0370] — Satterthwaite adjusted df = 165
Statistical Analysis 4: Comparison: Control Site - Rural Setting; Test type: Superiority or Other; p = .1555, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -.2564, 95% CI 2-sided [-.6086 to .0958] — Satterthwaite adjusted df = 157

6. Primary Outcome: Communication Satisfaction Questionnaire
Description: Communication satisfaction was measured utilizing a modified version of a 19-item measure of communication patterns between physicians and their clients (Campbell et al., 2007). Thirteen items focusing on the client's satisfaction with communication with their provider and their engagement in treatment were measured on a 7-point scale (strongly agree, agree, agree somewhat, undecided, disagree somewhat, disagree, strongly disagree). Example items included "My provider checks to be sure that I understand everything" or "My provider involves me in decisions as much as I want." Total average scores range from 1 to 7 with higher scores indicating better communication satisfaction. Analyses will examine change in Satisfaction Questionnaire scores from pre- to post-intervention.
Time Frame: Change in scores on the Communication Satisfaction Questionnaire from Baseline to 24 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Site - Urban Setting | Control Site - Urban Setting | Intervention Site - Rural Setting | Control Site - Rural Setting
Number analyzed (Participants) | 60 | 60 | 60 | 60
units on a scale
  Baseline: number analyzed (Participants) | 45 | 53 | 60 | 60
  Baseline | 4.283 (0.530) | 4.024 (0.706) | 4.363 (0.564) | 4.473 (0.578)
  24 Month Follow-up: number analyzed (Participants) | 30 | 39 | 34 | 46
  24 Month Follow-up | 3.947 (0.478) | 4.093 (0.529) | 4.135 (.769) | 4.065 (.690)
Statistical Analysis 1: Comparison: Intervention Site - Urban Setting; Test type: Superiority or Other; p = .0283, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -.2967, 95% CI 2-sided [-.5599 to -.0335] — Satterthwaite adjusted df = 213
Statistical Analysis 2: Comparison: Control Site - Urban Setting; Test type: Superiority or Other; p = .7407, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = .0401, 95% CI 2-sided [-.1969 to .2771] — Satterthwaite adjusted df = 194
Statistical Analysis 3: Comparison: Intervention Site - Rural Setting; Test type: Superiority or Other; p = .0619, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -.2338, 95% CI 2-sided [-.4778 to .0102] — Satterthwaite adjusted df = 186
Statistical Analysis 4: Comparison: Control Site - Rural Setting; Test type: Superiority or Other; p = .0009, Mixed Models Analysis — a priori test; Least Squares Mean Difference Test using LSMEANS pdiff test in SAS PROC MIXED 9.4; Mean Difference (Net) = -.3793, 95% CI 2-sided [-.5990 to -.1596] — Satterthwaite adjusted df = 172

ADVERSE EVENTS:
Time Frame: Every 6 months up to two years.
Description: Every 6 months, up to two years, research data (including information about adverse events) was collected. Serious adverse events (including death) were reported to the IRB.
Arm/Group | Intervention Site - Urban Setting | Control Site - Urban Setting | Intervention Site - Rural Setting | Control Site - Rural Setting
Serious Adverse Events (participants affected / at risk) | 3/60 | 5/60 | 1/60 | 1/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Site - Urban Setting (N=60) | Control Site - Urban Setting (N=60) | Intervention Site - Rural Setting (N=60) | Control Site - Rural Setting (N=60)
Serious Adverse Event (Death) (General disorders) | 3 (3) | 5 (5) | 1 (1) | 1 (1) — Cause of death was not related to the study's intervention.

LIMITATIONS AND CAVEATS:
Missing responses at baseline and 24 month followups were handled using full-information ML as part of a 2(Tx)x2(Location)x5(Time) mixed-effects ANOVA estimated using SAS PROC MIXED 9.4.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes